CLINICAL TRIAL: NCT00965471
Title: Effect of Chinese Traditional Medicine for Post Revascularization Treatment of Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Chinese Medicine (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other); Guangdong Provincial People's Hospital (Other); China-Japan Friendship Hospital (Other); Traditional Chinese Medicine Hospital of Xinjiang Uygur Autonomous Region (Unknown); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Teaching Hospital of Nanjin University of Traditional Chinese Medicine (Unknown); Second People's Hospital, Fujian Province (Other); Liaoning University of Traditional Chinese Medicine (Other); Guangzhou Overseas Chinese Hospital (Unknown); Beijing Tongren Hospital (Other); Shanghai 10th People's Hospital (Other); PLA.The Military General Hospital of Beijing (Unknown); The Sixth Affliated Hospital of Jinan University (Unknown); Beijing Anzhen Hospital (Other); Gansu Provincial Hospital (Other); Shaanxi Provincial People's Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); The Fifth Affliated Hospital of Guangxi Medical University (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006BAI04A01
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Percutaneous Coronary Artery Intervention; Coronary Artery Bypass Graft; Acute Coronary Syndrome
Keywords: percutaneous coronary artery intervention; coronary artery bypass graft; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- managed group (Experimental)
  Interventions: Drug: cipher prescription 1
- control group (Placebo Comparator)
  Interventions: Drug: cipher prescription 2

INTERVENTIONS:
Drug: cipher prescription 1 — Drug granules include ginseng,RADIX NOTOGINSENG,prepared RHIZOMA PINELLIAE with alumen radix glyrrhigae calcaren once daily for 180 days
  Arms: managed group
Drug: cipher prescription 2 — Placebo include amidon、bitter principles and diluents bases once daily for 180 days
  Arms: control group

SUMMARY:
The purpose of this study is to built the standard of Chinese Traditional Medicine test for Post percutaneous coronary artery intervention and coronary artery bypass graft，also for acute coronary syndrome，according to the multi-site、random large sample test.

ELIGIBILITY:
Inclusion Criteria:

* age40～75
* angina or CAD patient
* deficiency of heart-QI and blockage of phlegm and blood stasis in chinese medicine
* 1 week after operation，or 1week after drainage tube extraction for CABG
* sign a informed consent

Exclusion Criteria:

* severe cardia failure
* severe renal inadequacy
* complicating with malignant tumor,reactive alimentary tract hemorrhage and haematological systemic disorder etc.
* psychotic
* pregnant,lactation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
dead | 180±3days

SECONDARY OUTCOMES:
cardiovascular event | 180±3days

CONTACTS AND LOCATIONS:
Overall Officials: Ruan Xinmin, Study Chair — Guangzhou University of Chinese Medecine

REFERENCES:
- [Derived] Lin Y, Wang YF, Lin DQ, Chen JW, Li JZ, Lan TH, Ou AH, Ruan XM. Efficacy and safety of Huxin formula in patients after CABG: a multicenter, double-blind, randomized clinical trial. Forsch Komplementmed. 2014;21(6):351-9. doi: 10.1159/000370010. Epub 2014 Dec 11. PMID 25592946